CLINICAL TRIAL: NCT01243242
Title: Randomized, Double-blind, Placebo-controlled, Multi-center Study Designed to Evaluate the Efficacy, Safety and Tolerability of Metadoxine Extended Release in Adults With Attention Deficit Hyperactive Disorder
Brief Title: Clinical Efficacy & Safety, of Metadoxine (MG01CI) Extended Release in Attention-Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcobra Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AL008
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Results first posted 2012-04-18 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: ADHD
Keywords: ADHD,Adults,MG01CI,METADOXINE
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — metadoxine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- METADOXINE (Experimental): Eligible subjects will be randomly assigned to receive MG01CI (1,400 mg)
  Interventions: Drug: Metadoxine (MG01CI)
- Placebo (Placebo Comparator): Eligible subjects will be randomly assigned to receive Placebo (1,400 mg)
  Interventions: Drug: Metadoxine (MG01CI)

INTERVENTIONS:
Drug: Metadoxine (MG01CI) — MG01CI 1400 mg, that will be taken daily by the patients for a duration of 6 weeks.
  Other Names: Metadoxil

SUMMARY:
The purpose of this study is to evaluate efficacy, safety and tolerability of metadoxine (MG01CI) extended release formulation for the treatment of adults diagnosed with ADHD

DETAILED DESCRIPTION:
This will be a randomized, double-blind, placebo-controlled, parallel-group, multicenter study in adult subjects with ADHD.

Eligible subjects will be randomly assigned in a 1:1 ratio to one of two treatment groups, 1400 mg Metadoxine (MG01CI) and Placebo. The study will consist of three periods: a screening period of up to 2 weeks, a 6-week double-blind treatment period, and a 2-week safety follow-up period. The total duration of subject participation will be ~10 weeks.

Overview of Study Visits

Screening Period:

Visit 1 - Screening/Baseline Visit (up to 14 days prior to dosing)

Treatment Period:

Visit 2 - Day 0 (Randomization Visit) Visit 3 - Day 7 ± 2 days Visit 4 - Day 14 ± 2 days Visit 5 - Day 28 ± 2 days Visit 6 - Day 42 ± 2 days

Follow-up period:

Visit 7 - Day 56 ± 3 days

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females, 18 to 50 years old, inclusive, at screening visit
2. Diagnosed with ADHD based on

   1. DSM-IV criteria for ADHD as assessed by the Adult ADHD Clinician Diagnostic Scale (ACDS V1.2)
   2. SCID clinical interview
3. Clinical severity of at least a moderate level (Clinical Global Impression score of 4 or above)
4. Female subjects with childbearing potential must agree to use effective contraceptive and have negative urine pregnancy test at screening visit
5. Able to attend the clinic regularly and reliably
6. Able to swallow tablets/capsules
7. Able to understand, read, write and speak Hebrew fluently to complete study related materials
8. Able to understand and sign written informed consent to participate in the study

Exclusion Criteria:

1. Subjects who were non-responder to at least two ADHD treatments
2. Subjects with any medical or psychiatric condition (e.g. schizophrenia, personality disorder as diagnosed by DSM-IV) or clinical significant or unstable medical or surgical condition that may preclude safe and complete study participation as determined by medical history, physical examination, neurological exam, laboratory tests or ECG or based on the opinion of the Investigator; common diseases such as hypertension, type 2 diabetes mellitus, hyperlipidemia, etc. are allowed per the Investigator's judgment, as long as they are stable and controlled by medical therapy that is constant for at least 8 weeks prior to randomization and throughout the study
3. Any prescription or non-prescription ADHD medications during the 7 days prior to the screening visit
4. Known or suspected HIV-positive or with advanced diseases such as AIDS, Hepatitis C, Hepatitis B or tuberculosis
5. History of allergy or sensitivity to B complex vitamins
6. History or suspicion of PDD, NLD or other psychotic conditions
7. Use of Vitamin B throughout the study
8. Use of ADHD medications throughout the study
9. Use of any psychiatric medications throughout the study
10. Use of investigational medication/treatment in the past 30 days prior to the screening visit per the discretion of the Investigator
11. Use of any medication or food supplement not considered acceptable by the clinical Investigator or the medical monitor during the 14-day period before randomization
12. Current (or history within the last 6 months) of drug dependence or substance abuse disorder according to DSM-IV-TR criteria (excluding nicotine). Subjects should also agree to refrain from consuming abnormally high amounts of caffeine during the study.
13. Suicidality, defined as either active suicidal plan/intent or active suicidal thoughts, in the 6 months before the Screening Visit or no lifetime suicide attempt.
14. Blind subjects
15. Any relation to the Sponsor, Investigator or study staff
16. Any condition, which in the opinion of the Principal Investigator would place the subject at risk or influence the conduct of the study or interpretation of results, including (but not limited to) abnormally low intellectual capacity.
17. Subjects who cannot fully comprehend the implications of the protocol or comply with its requirements or are capable to follow the study schedule for any reason
18. Pregnancy, lactation or inadequate contraceptive method

    -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iris Manor, MD, Principal Investigator — Geha MC, Israel
Locations (2):
- Israel (2):
  - Cognitive Neurology unit Rambam Health Care Campus, Haifa
  - ADHD Unit, Geha Mental Health Center, Petah Tikva

REFERENCES:
- [Derived] Manor I, Newcorn JH, Faraone SV, Adler LA. Efficacy of metadoxine extended release in patients with predominantly inattentive subtype attention-deficit/hyperactivity disorder. Postgrad Med. 2013 Jul;125(4):181-90. doi: 10.3810/pgm.2013.07.2689. PMID 23933905
- [Derived] Manor I, Ben-Hayun R, Aharon-Peretz J, Salomy D, Weizman A, Daniely Y, Megiddo D, Newcorn JH, Biederman J, Adler LA. A randomized, double-blind, placebo-controlled, multicenter study evaluating the efficacy, safety, and tolerability of extended-release metadoxine in adults with attention-deficit/hyperactivity disorder. J Clin Psychiatry. 2012 Dec;73(12):1517-23. doi: 10.4088/JCP.12m07767. PMID 23290324

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects recruitment was done in two medical centers Geha and Rambam during Feb 2011-June 2011.
Pre-assignment Details: subjects were screened for study eligibility according to the inclusion exclusion criteria. Each subject underwent a battery of rating scales including confirmation of ADHD diagnosis and exclusion of other psychological disorders.In addition medical history was checked and lab test and Electrocardiogram (ECG) were preformed.
Groups:
- METADOXINE(MG01CI): Eligible subjects who received 1400 mg of Metadoxine
- Placebo: Eligible subjects who received 1400 mg of Placebo
Period: Overall Study
Arm/Group | METADOXINE(MG01CI) | Placebo
Started | 60 | 60
Completed | 57 | 56
Not Completed | 3 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 0 | 1
Not completed — sponsor decision | 0 | 1
Not completed — non compliance | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | METADOXINE(MG01CI) | Placebo | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 60 | 120
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 21 | 47
  Male | 34 | 39 | 73
Region of Enrollment [Number; unit: participants]
  Israel | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Conners' Adult ADHD Rating Scales (CAARS™)
Description: The primary efficacy endpoint is the difference in change (decrease) in CAARS (Total ADHD Symptoms Score) between the study groups. The CAARS assess the presence and severity of ADHD symptoms and behaviors in adults. Respondents are asked to report their own experiences by rating items pertaining to their behavior/problems using a 4-point Likert-style format ranging from 0 ('Not at all', 'never') to 3 ('Very much', 'very frequently'). The scale measures ADHD symptoms using a 30-item questionnaire.Total score is the sum of all the items ,min=30 Max=90
Time Frame: 6 weeks (from visit 1 baseline to visit 6)
Population: The ITT population included all randomized subjects who completed at least one post-randomization visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | METADOXINE(MG01CI) | Placebo
Number analyzed (Participants) | 58 | 59
units on a scale | -12 (9.69) | -8.93 (9.26)
Statistical Analysis 1: Comparison: METADOXINE(MG01CI) vs Placebo; For the primary endpoint (CAARS change), median test was applied as the primary analysis due to outlier numbers observed ; secondary analysis of the primary endpoint utilized ANCOVA with adjustment to age, gender and site (which is usually expected to influence the endpoint) as well as baseline values. Additional parametric T-test was applied, but was found less effective due to outlier values; Test type: Superiority or Other; p = 0.0093, Median — p value for the difference between groups in change from Screening to Termination was calculated using the median test for independent samples

2. Secondary Outcome: Test of Variables of Attention (TOVA) (Change in ADHD Score From Screening to Visit 6)
Description: The TOVA is a computerized test that provides information about an individual's sustained attention, speed and consistency of responding, and behavioral self-regulation and executive functioning. ADHD score is a comparison of the subject's response to the CPT test to those of an ADHD group, and is reported as a Z-score. An ADHD score of -1.80 and less fits the profile of the ADHD sample. A score of more than -1.80 (more positive) does not fit the ADHD profile. When comparing ADHD scores the higher the ADHD score the better the performance.
Time Frame: 6 weeks( visit 1 baseline to visit 6)
Population: The ITT population included all randomized subjects who completed at least one post-randomization visit.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | METADOXINE(MG01CI) | Placebo
Number analyzed (Participants) | 58 | 59
Z score | 4.96 (8.86) | 3.01 (6.40)
Statistical Analysis 1: Comparison: METADOXINE(MG01CI) vs Placebo; Analysis of Covariance (ANCOVA) was applied for comparing the differences in changes from screening/baseline (Visit 1) to termination (Visit 6) and to Visits 3 through 5 in the primary endpoint, CAARS, and secondary endpoint scales, CGI-S, TOVA and AAQoL between the study groups with adjustment to confounders (baseline score, site, age, gender, dose and past exposure to any other ADHD drug); Test type: Superiority or Other; p = 0.0195, ANCOVA — p value for the difference between groups in change from Screening to Termination was calculated using ANCOVA, adjusted for baseline score, gender, site and age

3. Secondary Outcome: Adult ADHD Quality of Life (AAQoL)- Measuring Change in Total Score of AAQoL From Visit 1 to Visit 6
Description: The AAQoL scale provides a validated disease-specific measure of the impact of ADHD on quality of life.It is scored as an overall score (29 items) and four subscale scores: life productivity (11 items), psychological health (6 items), life outlook (7 items) and relationships (5 items). Individual items are scored on a five-point Likert-like scale from 'Not at all/Never' (1) to 'Extremely/Very Often' (5).
Time Frame: 6 weeks (from visit 1 baseline to visit 6)
Population: The ITT population included all randomized subjects who completed at least one post-randomization visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | METADOXINE(MG01CI) | Placebo
Number analyzed (Participants) | 58 | 59
units on a scale | 10.93 (11.1) | 5.71 (15.82)
Statistical Analysis 1: Comparison: METADOXINE(MG01CI); Analysis of covariance (ANCOVA) was applied for comparing the differences in changes from screening/baseline (Visit 1) to termination (Visit 6) between the study groups with adjustment to confounders (baseline score, site, age, gender, dose and past exposure to any other ADHD drug); Test type: Superiority or Other; p = 0.0093, ANCOVA — [p-value comment as in outcome 2, analysis 1]

4. Secondary Outcome: Clinical Global Impression Scale (CGI-I)Score
Description: The CGI is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients). CGI-I scores range from 1 ('very much improved') through to 7 ('very much worse').
  During the conduct of the study, CGI-I evaluations were not done correctly and thus data interpretation is limited.
Time Frame: 6 weeks from visit 1 baseline to visit 6
Population: The ITT population included all randomized subjects who completed at least one post-randomization visit.
  During the conduct of the study, CGI-I evaluations were not done correctly and thus data interpretation is limited.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | METADOXINE(MG01CI) | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks (from time of informed consent to end of study)
Arm/Group | METADOXINE(MG01CI) | Placebo
Serious Adverse Events (participants affected / at risk) | 1/58 | 0/59
Other Adverse Events (participants affected / at risk) | 44/58 | 41/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | METADOXINE(MG01CI) (N=58) | Placebo (N=59)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | METADOXINE(MG01CI) (N=58) | Placebo (N=59)
Abdominal pain upper (Gastrointestinal disorders) | 5 (6) | 3 (3)
Asthenia (General disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Bacteriuria (Infections and infestations) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Disturbance in attention (Psychiatric disorders) | 2 (4) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (4) | 4 (5)
Fatigue (General disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 17 (22) | 23 (24)
Impatience (Psychiatric disorders) | 2 (2) | 0 (0)
Initial insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Memory impairment (Nervous system disorders) | 2 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (13) | 0 (0)
Nervousness (Psychiatric disorders) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (5)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less